CLINICAL TRIAL: NCT06035757
Title: The Effect of Administration of Sugammadex on the Occurrence of Emergence Agitation in Pediatric Strabismus Surgery-prospective Randomized Controlled Trial
Brief Title: The Occurrence of Emergence Agitation in Pediatric Strabismus Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Yea-Ji Lee, Assisstant professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KUMC2023-05-082
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Emergence Delirium; Strabismus; Pediatric ALL
MeSH Terms: conditions — Emergence Delirium; Strabismus; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Sugammadex; Injections; Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group pyridostigmine (Active Comparator): If TOF count is 1 or less, wait until it becomes 2 and then give the patient pyridostigmine dose of 350mcg/kg. If TOF count shows 4 with fade, 350mcg/kg of pyridostigmine is administered and without fade, 200mcg/kg is administered.
  Interventions: Drug: Pyridostigmine Bromide 5 MG/ML
- group sugammadex (Active Comparator): If TOF count shows 0 and PTC (posttetanic count) is 1 or more, sugammadex administered dose of 4mg/kg. If TOF count shows 1 or more, 2mg/kg is administered.
  Interventions: Drug: Bridion 200 MG in 2 ML Injection

INTERVENTIONS:
Drug: Bridion 200 MG in 2 ML Injection — Sugammadex is administered at the end of surgery after assessment of the level of neuromuscular blockade is done. The dosage of each reversal agent is determined with response to TOF or PTC.
  Other Names: Sugammadex
  Arms: group sugammadex
Drug: Pyridostigmine Bromide 5 MG/ML — Pyridostigmine is administered at the end of surgery after assessment of the level of neuromuscular blockade is done. The dosage of each reversal agent is determined with response to TOF.
  Other Names: Pyridostigmine
  Arms: group pyridostigmine

SUMMARY:
The present trial conducted to demonstrate the administration of sugammadex as reversal of neuromuscular blockade agent reduces the incidence of emergence agitation (EA) comparing to neostigmine

DETAILED DESCRIPTION:
EA is one of the most common postoperative complications in after general anesthesia in pre-school aged pediatric patients. There are several causes contributed to occurrence of EA such as postoperative pain, type of surgery and surgical site, hyperthermia or hypothermia. Some researches showed that the occurrence of EA is associated with patients' anxiety and investigators of this trial inferred that patients' anxiety after general anesthesia could be related to ability to breathe. Ability to breathe is highly associated with level of residual neuromuscular blockade (NMB) after recovery from general anesthesia. Investigators evaluate the Pediatric Anesthesia Emergence Delirium (PAED) Scale to investigate whether sugammadex as reversal agents of NMB reduces the incidence of EA in pediatric patients who undergo strabismus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled elective strabismus surgery aged 4-7 with American Society of Anesthesiologists (ASA) classification 1-3.

Exclusion Criteria:

* ASA classification 3 or more
* impaired liver function
* impaired kidney function
* myasthenia gravis or other neuromuscular disorders
* history of drug allergy
* cardiovascular disease or arrhythmia

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of EA in postanesthesia care unit (PACU) | EA is assessed three times at 15-minute intervals in PACU until discharge from PACU.
  EA is assessed with the PAED scale in PACU. EA is defined as the score is 10 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ji Lee, M.D Ph. D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul-T'ǔkpyǒlshi, South Korea